CLINICAL TRIAL: NCT07175727
Title: Safety and Efficacy of New, Non-thermal Ablation Techniques for the Treatment of Atrial Fibrillation - A Comparison of Two Ablation Systems
Brief Title: TWOSOME Trial: Single-Shot Versus Single-Tip Pulsed Field Ablation for Pulmonary Vein Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfried Krupp Krankenhaus (Other)
Responsible Party: Principal Investigator, Kars Neven, MD, PhD., Alfried Krupp Krankenhaus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 224/2022
Record Dates: First submitted 2025-08-28; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation (Paroxysmal)
Keywords: Pulsed Field Ablation; Pulmonary Vein Isolation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Single-Shot Pulsed Field Ablation (Active Comparator): Single-Shot Pulsed Field Ablation is performed using the FARAPULSE PFA System
  Interventions: Device: Pulmonary vein isolation; Radiation: cerebral magnetic resonance tomography; Diagnostic Test: Biomarker assessment (C-reacitve Protein, troponine)
- Single-Tip Pulsed Field Ablation (Active Comparator): Single-Tip Pulsed Field Ablation is performed using a conventional ablation catheter in combination with a pulsed field ablation generator.
  Interventions: Device: Pulmonary vein isolation; Radiation: cerebral magnetic resonance tomography; Diagnostic Test: Biomarker assessment (C-reacitve Protein, troponine)

INTERVENTIONS:
Device: Pulmonary vein isolation — Pulmonary vein isolation for paroxysmal atrial fibrillation
Radiation: cerebral magnetic resonance tomography — A subset of consecutive patients of each group (n=25 of each group) receives cMRI on the day after the procedure to asses silent cerebral lesions. A control cMRI is scheduled in case of positive findings.
Diagnostic Test: Biomarker assessment (C-reacitve Protein, troponine) — A subset of patients of each group (n=25 of each group) received blood tests to asses inflammation and troponine release.

SUMMARY:
Two non-thermal ablation techniques approved for routine clinical practice (CE-marked) for the interventional treatment of atrial fibrillation are compared in a 1:1 randomization to investigate patient data, procedural data, effectiveness, and safety.

DETAILED DESCRIPTION:
Patients with paroxysmal atrial fibrillation were randomized 1:1 to undergo pulmonary vein isolation using pulsed field ablation (PFA) with either single-shot PFA (FARAPULSE) or single-tip PFA (Galvanize Therapeutics). Baseline characteristics, procedural data, effectiveness, and safety outcomes were analyzed. In each group, a subset of consecutive patients underwent cerebral magnetic resonance imaging to assess silent cerebral lesions and was scheduled for biomarker assessment (blood sampling) to evaluate inflammation and troponin release after PFA.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent, symptomatic paroxysmal atrial fibrillation
* Age > 18 years
* Patient consen

Exclusion Criteria:

* Refusal of the patient
* Inability to provide informed consent
* Life expectancy < 2 years
* Pregnancy and breastfeeding (due to radiation exposure)
* History of left atrial ablation
* Known macro-reentry or focal atrial tachycardia
* Significant mitral valve stenosis
* History of heart valve replacement or reconstruction
* NYHA class III and IV
* Left ventricular ejection fraction < 35%
* Left atrial enlargement > 55 mm on echocardiography
* Intracardiac thrombus prior to the procedure
* Severe pulmonary disease with abnormal blood gases or requiring oxygen therapy
* Renal insufficiency (GFR < 30 mL/min) due to contrast medium use
* Stroke or TIA within the last 6 months
* Symptomatic carotid stenosis
* Active malignancy within the previous 24 months
* Untreated or uncontrolled thyroid disease
* Active bleeding or chronic bleeding tendency not amenable to curative treatment
* Body mass index > 35 kg/m²
* Contraindication to CT examination (e.g., contrast medium allergy or severe claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Freedom from arrhythmia | 12 months follow-up
  The clinical efficacy, e.g. freedom from atrial arrhythmias / atrial fibrillation is assessed by 5-7 day Holter Monitoring at 3, 6 and 12 months after the procedure. Any documented arrhythmia episode lasting >30s was calculated as failure. A three months blanking period was considered.

SECONDARY OUTCOMES:
Secondary outcomes: Complications, Silent cerebral lesions (cMRI) and biomarker assessments | 6 weeks
  All peri-procedural complications were noted. In a subset of consecutive patients (n = 25 in each group), cerebral magnetic resonance tomography (cMRI) was performed on the day after the ablation procedure to assess silent cerebral lesions. In case of positive cMRI findings (e.g. silent lesion), repeat cMRI was scheduled in 6 weeks. Biomarker analyses were performed using blood samples, e.g. high-sensitive troponin release at 6, 24 and 48 hours after the ablation as a marker of myocardial injury and C-reactive proteine levels before and 24 hours after the ablation procedure to asses inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Kars Neven, MD, PhD, Principal Investigator — Alfried Krupp Hospital; Stefan Hartl, Study Director — Alfried Krupp Hospital
Locations (1):
- Alfried Krupp Hospital, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after publication